CLINICAL TRIAL: NCT01612975
Title: The Effect of Perioperative Non-Steroidal Anti-Inflammatory Drug Naproxen on Pleural Effusion Formation After Lung Resection
Brief Title: The Effect of Non-Steroidal Anti-Inflammatory Drug Naproxen on Pleural Effusion Formation After Lung Resection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment futile
Sponsor: McMaster University (Other)
Collaborators: McMaster Surgical Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJHHNaproxenRCT
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2016-09

CONDITIONS: Pleural Effusion; Pleural Effusion Malignant
Keywords: Chest tubes; Length of stay; Pleural effusion; Lung resection; Post-operative; Lung cancer
MeSH Terms: conditions — Pleural Effusion; Pleural Effusion, Malignant; Lung Neoplasms | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): This study arm will encompass the administration of a placebo (physically identical to Naproxen) orally to participants. Naproxen is a painkiller with intrinsic anti-inflammatory properties, while the placebo has no pharmacological properties associated with it. Participants will also be taking Pantoprazole to negate the gastrointestinal consequences of Naproxen (or the placebo). Participants will not know which arm of the study they belong to. In addition, they will attend scheduled check-ups where their vitals will be recorded, as well as laboratory indicators of gastrointestinal complications (creatinine levels, etc) for their safety.
  Interventions: Drug: Placebo
- Naproxen (Experimental): Intervention arm involves administering 500mg Naproxen twice a day to participants and 40mg of Pantoprazole once a day in tandem. Pantoprazole will negate gastrointestinal consequences of Naproxen and reduce the likelihood of a complication occurring. Participants will take Naproxen at the above dosage from the time of surgery to four weeks following surgery. They will attend scheduled check-ups where their vitals will be recorded, as well as laboratory indicators of gastrointestinal complications (creatinine levels, etc) for their safety. This experiment is double-blinded so neither investigators nor participants will know which arm of the study they belong to.
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: Naproxen — Intervention arm involves administering 500mg Naproxen BID to participants and 40mg of Pantoprazole in tandem. Pantoprazole will negate gastrointestinal consequences of Naproxen and reduce the likelihood of a complication occurring. Participants will take Naproxen at the above dosage from the time of surgery to four weeks following surgery. They will attend scheduled check-ups where their vitals will be recorded, as well as laboratory indicators of gastrointestinal complications (creatinine levels, etc) for their safety. This experiment is double-blinded so neither investigators nor participants will know which arm of the study they belong to.
  Arms: Naproxen
Drug: Placebo — Inert, inactive placebo pill similar in appearance to naproxen allocation. To be taken twice daily for 4 weeks total along with 40mg pantoprazole.
  Arms: Placebo

SUMMARY:
Following a lung resection procedure, patients have their pleural space drained of fluid that accumulates due to the severing of proximal vessels like lymph nodes. The volume of fluid pumped depends on the severity of the inflammation. The investigators are conduction this study to attempt to use painkillers with intrinsic anti-inflammatory action to try and reduce the degree of inflammation in patients' pleural cavity, thus ensuring patients are discharged faster, with a greater comfort level, and a hopefully lower rate of admission.

DETAILED DESCRIPTION:
In this study the investigators will attempt to reduce the degree of inflammation (and thus polymorphonuclear leukocyte counts) in the pleural space following a lung resection procedure by administering the Non Steroid Anti-Inflammatory Drug (NSAID) Naproxen in tandem with Proton Pump Inhibitor (PPI) Pantoprazole, ideally leading towards a significantly reduced volume of transudate and exudate generated.

This will be achieved by running a placebo-controlled double blinded randomized control trial where investigators and participants will be blinded so as to eliminate experimenter bias. After screening for suitable participants using stringent inclusion and exclusion criteria, patients will be administered by allied health professionals 500mg Naproxen twice daily and 40mg Pantoprazole once daily, or an identical placebo for four weeks following resection surgery. Patients will undergo a thorough examination during their scheduled follow-up appointments to monitor general vitals as well as possible gastrointestinal complications. The primary outcome is a significant reduction (Δ100ml) of chest fluid extracted in the intervention arm of the study in comparison to that of the control arm. Secondary outcomes will include a reduction in length of stay measured in days between control and intervention arms as well as a reduction in the total number of days chest tubes are retained in-situ. Conditions such as mortality and morbidity, the onset of complications, and general re-admission rates will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older
* Participants must be undergoing a major lung resection due to primary or secondary malignancy
* Must have an aptitude for following directions and commitment to the study

Exclusion Criteria:

* Patients who are unable to read and communicate in English
* Patients undergoing a pneumonectomy or Open lung resection
* Previous treatments on the same anatomical side including chemotherapy, radiation therapy, and radio-frequency ablation
* Patients who have undergone decortication for empyema or malignancy.
* Patients who have a chest tube in-situ for persistent air leak
* Patients with clinical or laboratory indicators of renal failure, defined as serum creatinine level of 170µmol/l
* Patients with active or previous history of peptic ulcer disease
* Patients with a known intolerance to Proton Pump Inhibitors (PPIs)
* Known allergy to study drugs
* Use of NSAIDs 4 weeks prior to randomization or on-going use of NSAIDs.
* The use of any medications known to reduce inflammation, including but not limited to: steroids (both oral and intravenously), methotrexate, COX-II inhibitors, other NSAIDs
* Chest tube for persistent air leak.
* Patients who are pregnant or lactating
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-04; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in volume of pleural effusion collected | 4 weeks
  The investigators are looking to measure the volume of pleural effusion collected from in-situ chest tubes in patients following a lung resection, measured in mL

SECONDARY OUTCOMES:
Hospital length of stay; compared between intervention and control arms | 4 weeks
  The length of stay will be measured from the admitting day to the day of discharge to home.
Gastrointestinal complications | 4 weeks
  Recorded as a binary event, adverse events related to the gastrointestinal tract may occur in participants undergoing treatment. The extent of this occurrence will determine whether or not further intervention by the Data and Safety Monitoring Committee is necessary.
General re-admission rates | 4 weeks
  Participants recently discharged following a lung resection have a chance to be re-admitted for a post-operative complication. This will be measured as a binary event and the total associated length of stay associated with the episode.
Total number of days chest tubes remain in-situ | 4 weeks
  This outcome is related to the volume of pleural effusion produced and will measure the time chest tubes remain in place following surgery, measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Shargall, MD, BSc, FRCSC, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Watanabe A, Watanabe T, Ohsawa H, Mawatari T, Ichimiya Y, Takahashi N, Sato H, Abe T. Avoiding chest tube placement after video-assisted thoracoscopic wedge resection of the lung. Eur J Cardiothorac Surg. 2004 May;25(5):872-6. doi: 10.1016/j.ejcts.2004.01.041. PMID 15082297
- [Background] Cerfolio RJ, Bryant AS. Results of a prospective algorithm to remove chest tubes after pulmonary resection with high output. J Thorac Cardiovasc Surg. 2008 Feb;135(2):269-73. doi: 10.1016/j.jtcvs.2007.08.066. PMID 18242249
- [Background] Suemitsu R, Ondo K, Fukuyama S, Ueda H. Late-period-onset chylothorax after a pulmonary resection for lung cancer: a case report. Ann Thorac Cardiovasc Surg. 2007 Oct;13(5):345-8. PMID 17954994
- [Background] Kroegel C, Antony VB. Immunobiology of pleural inflammation: potential implications for pathogenesis, diagnosis and therapy. Eur Respir J. 1997 Oct;10(10):2411-8. doi: 10.1183/09031936.97.10102411. PMID 9387973
- [Background] Scheiman JM, Hindley CE. Strategies to optimize treatment with NSAIDs in patients at risk for gastrointestinal and cardiovascular adverse events. Clin Ther. 2010 Apr;32(4):667-77. doi: 10.1016/j.clinthera.2010.04.009. PMID 20435236
- [Background] Trelle S, Reichenbach S, Wandel S, Hildebrand P, Tschannen B, Villiger PM, Egger M, Juni P. Cardiovascular safety of non-steroidal anti-inflammatory drugs: network meta-analysis. BMJ. 2011 Jan 11;342:c7086. doi: 10.1136/bmj.c7086. PMID 21224324
- [Background] Ackerman N, Tomolonis A, Miram L, Kheifets J, Martinez S, Carter A. Three day pleural inflammation: a new model to detect drug effects on macrophage accumulation. J Pharmacol Exp Ther. 1980 Dec;215(3):588-95. PMID 7441518
- See also: Related Info — http://library.med.utah.edu/WebPath/INFLHTML/INFL062.html